CLINICAL TRIAL: NCT03099473
Title: A Randomized Trial of Ocular Electroacupuncture for Trochlear Nerve Palsy
Brief Title: Effects of Ocular Electroacupuncture on Trochlear Nerve Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017031602
Record Dates: First submitted 2017-03-24; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Trochlear Nerve Palsy
Keywords: electroacupuncture; trochlear nerve palsy; eyeball movement; diplopia; ocular motility disorder
MeSH Terms: conditions — Trochlear Nerve Diseases; Diplopia; Ocular Motility Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ocular electroacupuncture (Experimental): Patients will receive electroacupuncture for 40 mins with certain parameter at ocular area, once daily, 5 times a week and 6 weeks in all. The acupoints are selected based on the anatomy of extraocular muscles innervated by trochlear nerve.
  Interventions: Other: ocular electroacupuncture
- ocular acupuncture (Experimental): Patients will receive acupuncture for 40 mins at ocular area, once daily, 5 times a week and 6 weeks in all. The acupoints are selected based on the anatomy of extraocular muscles innervated by trochlear nerve.
  Interventions: Other: ocular acupuncture
- sham acupuncture (Sham Comparator): Patients will receive sham acupuncture for 40 mins at ocular area, once daily, 5 times a week and 6 weeks in all. The acupoints are selected based on the anatomy of extraocular muscles innervated by trochlear nerve. When the care provider performed operating acupuncture, the needles of sham acupuncture set will not be inserted into the skin of patient.
  Interventions: Other: sham acupuncture

INTERVENTIONS:
Other: ocular electroacupuncture — During intervention period, patients will continue to keep medications for primary condition. Patient's skin located in the extraocular muscles projection area is routinely disinfected. A diameter of 0.20 mm and length of 25 mm needle is inserted slowly. Piercing depth is about 20mm. The electropuncture apparatus is used, each group of electrodes are distinguished with different colors of wires to generate current stimulations of current 1.0~1.5 milliampere (mA), voltage 9 volt(V), frequency 1.5 hertz (Hz), and duration of 40 minutes.
  Arms: ocular electroacupuncture
Other: ocular acupuncture — During intervention period, patients will continue to keep medications for primary condition. Patient's skin located in the extraocular muscles projection area is routinely disinfected. A diameter of 0.20 mm and length of 25 mm needle is inserted slowly. Piercing depth is about 20mm.The duration of intervention is 40 minutes.
  Arms: ocular acupuncture
Other: sham acupuncture — During intervention period, patients will continue to keep medications for primary condition. Patient's skin located in the extraocular muscles projection area is routinely disinfected. A diameter of 0.20 mm and length of 25 mm sham needle set is stick onto insertion area without piercing into the skin. The duration of intervention is 40 minutes.
  Arms: sham acupuncture

SUMMARY:
The purpose of the study is to testify the efficacy of treating trochlear nerve palsy with ocular electroacupuncture or ocular acupuncture, and to compare the efficacy between these two interventions.

DETAILED DESCRIPTION:
The purpose of the study is to testify whether ocular electroacupuncture or ocular acupuncture is effective for trochlear nerve palsy (TNP), through treating TNP patient for 6 weeks, using self-invented acupoints according to anatomy of extraocular muscles innervated by trochlear nerve, and using sham acupuncture as controlled group, and try to provide clinical evidence for promoting these new techniques.

ELIGIBILITY:
Inclusion criteria;

1. patient with confirmed diagnosis of trochlear nerve palsy made by neurologist or ophthalmologist;
2. patient in stable condition after treatment for primary disease;
3. age between 18 to 80 years old without gender limitation;
4. haven't received acupuncture intervention for TNP before;
5. patient with conscious, willing to cooperate and voluntarily agreed to participate and signed informed consent forms.

Exclusion criteria:

1. those with other diagnosed medical conditions known to contribute to TNP symptoms, such as thyroid disease, myasthenia gravis, mitochondrial myopathy, congenital strabismus or received strabismus surgery;
2. those with color blindness, dyschromatopsia or abnormal retinal correspondence couldn't complete computerized diplopia test;
3. those with serious medical conditions that might limit their participation;
4. those with eye or other location with serious infections;
5. women who had a positive pregnancy test or who were planning to become pregnant during the study period;
6. those with bleeding tendency, blood coagulation dysfunction or taken anticoagulant drugs;
7. who had participate in other clinical trials, which may affect the results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-04-06 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Angle of diplopia deviation at 6 Weeks | 6 week
  Patients will receive computerized diplopia test with the guidance from an investigator. The data will be generated by the software automatically. The changes from baseline will be recorded.

SECONDARY OUTCOMES:
The quality of life questionnaire for ocular motor nerve palsy | 6 week
  The patients will finish a questionnaire to evaluate their physical and psychological status during this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Lingyun Zhou, PhD, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The first affiliated hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No